CLINICAL TRIAL: NCT01041508
Title: Phase I Feasibility Study of Clofarabine and Low Dose Total Body Irradiation (TBI) as a Non-myeloablative Preparative Regimen for Stem Cell Transplantation (SCT) for Hematologic Malignancies
Brief Title: Clofarabine and Low Dose Total Body Irradiation as a Preparative Regimen for Stem Cell Transplant in Leukemia.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Therapeutic Advances in Childhood Leukemia Consortium (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T2008-005; IND 101588 (Other: FDA); NCT00884572 (obsolete NCT alias)
Record Dates: First submitted 2009-12-29; First posted 2009-12-31 (Estimated); Results first posted 2024-02-01 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2023-05

CONDITIONS: Leukemia Lymphoblastic, Acute; Acute Myeloid Leukemia; Neoplasm Recurrent
Keywords: ALL; AML; Recurrence; Relapsed; Stem Cell Transplant; Non-myeloablative
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Recurrence | interventions — Clofarabine; Whole-Body Irradiation; Stem Cell Transplantation; Cyclosporine; Cyclosporins; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Related Donor Arm (Experimental): Patients with related stem cell donors. Patients will receive Clofarabine in combination with 2Gy total body irradiation (TBI) as a preparative regimen for stem cell transplantation, in turn followed by cyclosporine and Mycophenolate Mofetil as GVHD prophylaxis.
  Interventions: Drug: Clofarabine; Radiation: Total Body Irradiation; Other: Stem Cell Transplantation; Drug: Cyclosporine; Drug: Mycophenolate Mofetil
- Unrelated Donor Arm (Experimental): Patients with unrelated stem cell donors. Patients will receive Clofarabine in combination with 2Gy total body irradiation (TBI) as a preparative regimen for stem cell transplantation, in turn followed by cyclosporine and Mycophenolate Mofetil as GVHD prophylaxis.
  Interventions: Drug: Clofarabine; Radiation: Total Body Irradiation; Other: Stem Cell Transplantation; Drug: Cyclosporine; Drug: Mycophenolate Mofetil

INTERVENTIONS:
Drug: Clofarabine — Clofarabine will be given as an intravenous infusion over 2 hours on days -6 though -2. The dose of Clofarabine will be assigned at study entry (30, 40 or 52 mg/m2).
  Other Names: Clolar; Evoltra
Radiation: Total Body Irradiation — Low dose (2 Gy) TBI will be administered from a linear accelerator at ≤ 20 cGy/min on day "0" according to institutional guidelines.
  Other Names: TBI
Other: Stem Cell Transplantation — Patients will be infused with 'unmanipulated' hematopoietic stem cells from a related or unrelated donor on day 0 of the treatment regimen according to institutional practice guidelines.
  Other Names: SCT
Drug: Cyclosporine — Cyclosporine is given IV based on body weight at:
  * Age ≤ 6 years old: 6 mg/kg IV QD. in divided doses (e.g. 2 mg/kg q8hrs).
  * Age > 6 years old: 3 mg/kg IV QD in divided doses (1.5mg/kg q12hrs)
  Cyclosporine should be started on day -1 after completion of Clofarabine. Levels should be maintained between 300-400 ng/ml.
  Other Names: Gengraf; Neoral; Sandimmune
Drug: Mycophenolate Mofetil — MMF will be at 15 mg/kg, based on adjusted body weight, q 8 hours (45 mg/kg/day; max.3g/day) PO, or IV if indicated, from the evening of day 0 (i.e. first dose 4-6 hours following stem cell infusion) to day +40 post-transplant. Oral doses will be rounded to the nearest 250 mg (capsules are 250 mg). MMF is also available in oral suspension form. MMF will be given until day +40 post transplant and then tapered by 10% per week to be discontinued by day +90.
  Other Names: MMF

SUMMARY:
Stem cell transplant is an important therapeutic option for pediatric patients with relapsed or refractory leukemia. Although, full myeloablative transplants are widely used for patients with acute leukemia, myeloablative chemo-radiotherapy may not be feasible in some specific settings. These settings include 1) patients with pre-existing health issues and organ toxicities; 2) patients who have relapsed post-ablative transplant and need a second stem cell transplant; and 3) leukemia patients with advanced disease who have been heavily pre-treated. Clofarabine, a new purine nucleoside anti-metabolite, has the advantage of significant antileukemic activity in addition to its possible immuno-suppressive properties. In this study we plan to determine the maximum feasible dose (MFD) of Clofarabine in combination with total body irradiation that can achieve durable donor engraftment without causing excessive toxicity.

DETAILED DESCRIPTION:
Standard non-myeloablative regimens use Fludarabine and low dose total body irradiation (TBI) as pioneered by the Seattle group. Fludarabine is mainly used for its immuno-suppressive properties and has limited anti-leukemic effects. Since, the non-myeloablative and RIC regimens do not include intensive chemotherapy; relapse rates can be higher in RIC regimens compared to full myeloablative regimens. One way to improve overall survival in non-myeloablative / RIC setting is to add more effective anti-leukemia agents to prevent post-transplant relapses, without increasing TRM. Clofarabine, a new purine nucleoside anti-metabolite, has the advantage of significant antileukemic activity in addition to its possible immuno-suppressive properties. Combining Clofarabine with low dose TBI as a non-myeloablative preparative regimen may improve overall outcomes of SCT in advanced hematological malignancies. Therefore, in this study we plan to determine the maximum feasible dose (MFD) of Clofarabine in combination with 2Gy TBI that can achieve durable donor engraftment without causing excessive toxicity. The MFD determined from this pilot will be used in the next phase to study the outcomes after using this combination for SCT in this very high risk population.

ELIGIBILITY:
Inclusion Criteria

Since this is a Phase 1 study, any patient who is a candidate for a non-myeloablative SCT because he/she cannot tolerate the standard myeloablative preparative therapy is eligible for this trial. Briefly, the following groups of patients will be targeted and are eligible for this trial:

* Patients with presence of organ system dysfunction or severe systemic infections that significantly increase the risk of TRM with standard myeloablative regimens.
* History of previous myeloablative allogeneic or autologous transplantation.
* Heavily pre-treated leukemia patients, eg. Patients in CR after failure of ≥2 prior regimens.(eg. ALL CR ≥ 3).
* Combination of toxicities or co-morbidities that leads the investigator to feel that the child is at high risk (>50%) of TRM with standard ablative regimens.

The eligibility criteria listed below are interpreted literally and cannot be waived.

1. Age: Patients must be >1 and < 21 years of age at the of study entry.
2. Diagnosis

   1. Patients must have a diagnosis of ALL or AML.

      * ALL patients must be in clinical remission defined as BM morphology <5% blasts and CNS 1 status.
      * AML patients must be in M1 (<5% blasts) or M2 (<20% blasts) marrow status with CNS 1 status.
   2. Patient must have an ANC > 750/ul.
3. Donor Selection: Patient must have one of the appropriate donor types as described below:

   1. HLA identical sibling donor.
   2. Complete matched unrelated donor, (matched at A, B, C, DR B1 and DQ, B1 at the allelic level based on high resolution typing for Class I and II antigens, 10/10 match).
   3. 1 allelic mis-matched unrelated donor (antigen mis-matches are not allowed).
4. Stem Cell Source: The stem cell source from the donor must be one of the following:

   1. Bone Marrow or Peripheral blood stem cells (PBSC) from a matched related donor.
   2. PBSC from an unrelated donor. (Bone marrow is not acceptable for unrelated donors)
5. Performance Level: Karnofsky > 50% for patients > 10 years of age and Lansky > 50% for patients < 10 years of age.
6. Reproductive Function

   1. Female patients of childbearing potential must have a negative serum pregnancy test confirmed within 2 weeks prior to enrollment.
   2. Female patients with infants must agree not to breastfeed their infants while on this study.
   3. Male and female patients of child-bearing potential must agree to use an effective method of contraception approved by the investigator during the study.
7. Renal and Hepatic Function: Patient must have adequate renal and hepatic functions as indicated by the following laboratory values:

   1. Patients must have a calculated creatinine clearance ≥ 70mL/min/m2 as calculated by the Schwartz formula for estimated glomerular filtration rate (GFR) where GFR (ml/min/1.73 m2) = k * Height (cm)/serum creatinine (mg/dl). K is a proportionality constant which varies with age and is a function of urinary creatinine excretion per unit of body size; 0.45 up to 12 months of age; 0.55 children and adolescent girls; and 0.70 adolescent boys.
   2. Total serum bilirubin < 2 mg/dL.
   3. Aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 5 × ULN.
8. Cardiac Function: Patient must have a shortening fraction (SF) > 25%. If the SF is <25%, patient must have an ejection fraction (EF) by MUGA of >30%. 3.3.9 Pulmonary Function Patient must have pulmonary function as defined below:

   1. DLCO >30%
   2. FVC/TLC >30%
   3. FEV1 > 30% of predicted
   4. Patient is not on continuous oxygen

   If patient is not old enough or unable to comply with pulmonary function tests, they must have a pulse ox >92% in room air and not be on continuous oxygen.
9. Patients with prior exposure to Clofarabine are eligible.
10. Informed Consent: Patients and/or their parents or legal guardians must be capable of understanding the investigational nature, potential risks and benefits of the study. All patients and/or their parents or legal guardians must sign a written informed consent. Age appropriate assent will be obtained per institutional guidelines. To allow non-English speaking patients to participate in this study, bilingual health services will be provided in the appropriate language when feasible.
11. Protocol Approval: All institutional, FDA, and OHRP requirements for human studies must be met.

Exclusion Criteria

Patients will be excluded if they meet any of the following criteria:

1. Infection

   1. Patients will be excluded if they have evidence of an active, progressive invasive infection. All patients with existing infections at the time study entry should be discussed with the study chair.

      * Patients may have stable invasive infections and still be eligible.
      * Patients with infections that are responsive to medical or surgical treatment as shown by radiographic and or microbial assessment may still be eligible.
   2. Patients will be excluded if they have an active, uncontrolled systemic fungal, bacterial, viral or other infection. All patients with existing infections at the time of study entry should be discussed with the study chair.

      * An active uncontrolled infection is defined as exhibiting ongoing signs and symptoms related to the infection (fevers, positive blood cultures, chills, tachycardia, etc) despite appropriate antibiotics or other treatment.
2. Patient has a diagnosis of CML or MDS.
3. Patient has CNS 2 or CNS 3 status.
4. Patient is HIV positive.
5. Current or planned treatment with chemotherapy, radiation therapy, or immunotherapy other than as specified in the protocol.
6. Use of investigational agents within 30 days or any anticancer therapy within 2 weeks before study entry.
7. Have any other severe concurrent disease, or have a history of serious organ dysfunction or disease involving the heart, kidney (including dialysis patients), liver, or other organ system that may place the patient at undue risk to undergo treatment.
8. Patients with a systemic fungal, bacterial, viral, or other infection not controlled (defined as exhibiting ongoing signs/symptoms related to the infection and without improvement, despite appropriate antibiotics or other treatment).
9. Any significant concurrent disease, illness, psychiatric disorder or social issue that would compromise patient safety or compliance, study participation, follow up, or interpretation of study results.

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Actual)
Dates: Start 2010-01-29 (Actual); Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandeep Soni, MD, Study Chair — Nationwide Childrens Hospital; Haydar Frangoul, MD, Study Chair — Vanderbilt University
Locations (6):
- United States (6):
  - Childrens Hospital Los Angeles, Los Angeles, California
  - Nationwide Childrens Hospital, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Vanderbilt Children's Hospital, Nashville, Tennessee
  - Primary Children's Hospital, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington

REFERENCES:
- [Result] Soni S, Abdel-Azim H, McManus M, Nemecek E, Sposto R, Woolfrey A, Frangoul H. Phase I Study of Clofarabine and 2-Gy Total Body Irradiation as a Nonmyeloablative Preparative Regimen for Hematopoietic Stem Cell Transplantation in Pediatric Patients with Hematologic Malignancies: A Therapeutic Advances in Childhood Leukemia Consortium Study. Biol Blood Marrow Transplant. 2017 Jul;23(7):1134-1141. doi: 10.1016/j.bbmt.2017.03.037. Epub 2017 Apr 7. PMID 28396162
- See also: Therapeutic Advances in Childhood Leukemia & Lymphoma Consortium web site — http://www.tacl.us

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: At each dose level, after the first 3 patients or after 6 patients, the dose level will be either escalated to the next dose level, expanded, or de-escalated, or the study will be halted, depending on the number of observed Transplant Related Mortality (TRM) or Severe Renal Insufficiency (SRI) and Non-engraftment (NE) and evaluation status of surrounding dose levels.
Groups:
- Cohort A - Related Donor- Dose Level 1: Dose Level 1 Clofarabine 40 mg/m^2. Cohort A will include patients who have matched related donors.
- Cohort B - Related Donor- Dose Level 2: Dose Level 2 Clofarabine 52 mg/m^2. Cohort B will include patients who have matched related donors.
- Cohort C- Unrelated Donor- Dose Level 1: Dose Level 1 Clofarabine 40 mg/m^2. Cohort C will include patients who have unrelated donors.
- Cohort D- Unrelated Donors- Dose Level 2: Dose Level 2 Clofarabine 52 mg/m^2. Cohort D will include patients who have unrelated donors.
Period: Overall Study
Arm/Group | Cohort A - Related Donor- Dose Level 1 | Cohort B - Related Donor- Dose Level 2 | Cohort C- Unrelated Donor- Dose Level 1 | Cohort D- Unrelated Donors- Dose Level 2
Started | 3 | 6 | 3 | 6
Completed | 3 | 6 | 3 | 6
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participating subjects receiving the non-myeloablative preparative regimen followed by hematopoetic stem cell transplantation
Groups:
- Cohort A- Related Donor- Dose Level 1: Dose Level 1 Clofarabine 40 mg/m^2. Cohort A will include patients who have matched related donors.
- Cohort B- Related Donor - Dose Level 2: Dose Level 2 Clofarabine 52 mg/m^2. Cohort B will include patients who have matched related donors.
- Cohort C- Unrelated Donor - Dose Level 1: Dose Level 1 Clofarabine 40 mg/m^2. Cohort C will include patients who have matched unrelated donors.
- Cohort D- Unrelated Donor - Dose Level 2: Dose Level 2 Clofarabine 52 mg/m^2. Cohort D will include patients who have matched unrelated donors.
- Total: Total of all reporting groups
Arm/Group | Cohort A- Related Donor- Dose Level 1 | Cohort B- Related Donor - Dose Level 2 | Cohort C- Unrelated Donor - Dose Level 1 | Cohort D- Unrelated Donor - Dose Level 2 | Total
Number analyzed (Participants) | 3 | 6 | 3 | 6 | 18
Age, Continuous [Median (Full Range); unit: years] | 15 [8 to 15] | 5.5 [1 to 13] | 3.5 [3 to 10] | 9 [1 to 18] | 14.5 [3 to 18]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 1 | 3 | 10
  Male | 1 | 2 | 2 | 3 | 8
Diagnosis [Count of Participants; unit: Participants]
  Acute Lymphoblastic Leukemia (ALL) | 2 | 4 | 2 | 3 | 11
  Acute Myeloid Leukemia (AML) | 1 | 2 | 1 | 3 | 7
Prior myeloablative allogeneic HSCT [Count of Participants; unit: Participants] | 0 | 1 | 0 | 0 | 1
Prior liver transplantation [Count of Participants; unit: Participants] | 2 | 2 | 2 | 2 | 8
Trisomy 21 [Count of Participants; unit: Participants] | 3 | 3 | 3 | 3 | 12
Donor type [Count of Participants; unit: Participants]
  Related Donor | 3 | 6 | 0 | 0 | 9
  Unrelated Donor | 0 | 0 | 3 | 6 | 9
Stem cell source [Count of Participants; unit: Participants]
  Peripheral Blood | 3 | 3 | 3 | 6 | 15
  Bone Marrow | 0 | 3 | 0 | 0 | 3
CD34+ cell dose [Median (Full Range); unit: million cells per kg] | 6.8 [2.2 to 11.5] | 6.8 [2.2 to 11.5] | 6.8 [2.2 to 11.5] | 6.8 [2.2 to 11.5] | 6.8 [2.2 to 11.5]
Performance Status [Count of Participants; unit: Participants] — The Karnofsky Performance Scale Index allows patients to be classified as to their functional impairment. This can be used to compare effectiveness of different therapies and to assess the prognosis in individual patients. The lower the Karnofsky score, the worse the survival for most serious illnesses. The scale ranges from 0 to 100, with intervals divisible by 10. Each interval represents a pre-determined description of the patients ability to carry out everyday tasks and to take care of themselves. The patients is evaluated and assigned a scale score by a qualified healthcare professional.
  Participants
    90-100 | 1 | 4 | 3 | 5 | 13
    80-90 | 1 | 2 | 0 | 1 | 4
    50-80 | 1 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Maximum Feasible Dose of Clofarabine
Description: The primary objective of the study is to determine the maximum feasible dose (MFD) of Clofarabine that can be given in combination with 2Gy total body irradiation as a non-myeloablative preparative regimen for allogeneic stem cell transplantation in pediatric patients with relapsed leukemia. The MFD is defined as the highest clofarabine dose associated with both an acceptably low toxicity and low non-engraftment (NE) rate. NE is defined as < 5% donor T cells at any time point during serial monitoring. Monitoring during the evaluation period is required Day +30, +60 and +100.
Time Frame: Day +100
Population: This analysis was performed for the entire study population. Cohorts were not separately analyzed for the maximum feasible dose of clofarabine.
Measure: Number; unit: mg/m^2
Groups:
- Entire Study Population: Maximum Feasible Dose (MFD) was analyzed across all cohorts of the study. This includes all 18 patients who were enrolled on to this trial
Arm/Group | Entire Study Population
Number analyzed (Participants) | 18
mg/m^2 | 52

2. Secondary Outcome: Days of Engraftment in Both Matched Related Donor (MRD) and Matched Unrelated Donor (MUD)
Description: Donor engraftment will be assessed by serial monitoring of T-cell (CD3) and myeloid (CD33) chimerism at day +30, 60, 100, 180 and 1 year at the local institution using PCR based VNTR/STR amplification techniques. Neutrophil engraftment is defined as first day of an ANC ≥500/μL on 3 consecutive measurements.
Time Frame: Days +30, 60, 100, 180
Measure: Median (Full Range); unit: Days
Groups:
- Cohort A- Related Donor- Dose Level 1: Dose Level 1 is the starting dose level of Clofarabine will be 40 mg/m2/dose given day -6 through -2. A modified 3+3 patient cohort dose escalation and de-escalation design. Cohort A will include patients who have matched related donors.
- Cohort B- Related Donor- Dose Level 2: Dose Level 2 of Clofarabine will be administered 52 mg/m2/dose Day -6 through -2. Cohort B will include patients who have matched related donors.
- Cohort C- Unrelated Donor- Dose Level 1: Dose Level 1 is the starting dose level of Clofarabine will be 40 mg/m2/dose given day -6 through -2. A modified 3+3 patient cohort dose escalation and de-escalation design. Cohort C will include patients who have unrelated donors.
- Cohort D- Unrelated Donor- Dose Level 2: Dose Level 2 of Clofarabine will be administered 52 mg/m2/dose Day -6 through -2. Cohort D will include patients who have unrelated donors.
Arm/Group | Cohort A- Related Donor- Dose Level 1 | Cohort B- Related Donor- Dose Level 2 | Cohort C- Unrelated Donor- Dose Level 1 | Cohort D- Unrelated Donor- Dose Level 2
Number analyzed (Participants) | 3 | 6 | 3 | 6
Days | 20 [17 to 22] | 19.5 [14 to 25] | 19 [19 to 20] | 15.5 [9 to 19]

3. Secondary Outcome: Transplant Related Mortality (TRM) at Day +100
Description: TRM is defined as any mortality within the first 100 days post stem cell infusion associated with regimen related toxicity, infection, or GVHD.
Time Frame: Day 100
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A- Related Donor- Dose Level 1 | Cohort B- Related Donor- Dose Level 2 | Cohort C- Unrelated Donor- Dose Level 1 | Cohort D- Unrelated Donor- Dose Level 2
Number analyzed (Participants) | 3 | 6 | 3 | 6
Participants | 0 | 0 | 0 | 0

4. Secondary Outcome: Days to Platelet Recovery
Description: Platelet recovery is defined as the first day of 3 consecutive measurements of platelets ≥20,000/μL after at least 7 days without transfusion support.
Time Frame: Days +30, 60, 100, 180
Measure: Mean (Full Range); unit: Days
Arm/Group | Cohort A- Related Donor- Dose Level 1 | Cohort B- Related Donor- Dose Level 2 | Cohort C- Unrelated Donor- Dose Level 1 | Cohort D- Unrelated Donor- Dose Level 2
Number analyzed (Participants) | 3 | 6 | 3 | 6
Days | 10 [7 to 17] | 13.5 [3 to 29] | 11 [9 to 11] | 10.5 [6 to 16]

5. Post Hoc Outcome: Number of Participants With Acute GVHD ≥ Grade 2
Description: Acute GVHD was graded according to consensus grading criteria (Przepiorka D, Weisdorf D, Martin P, et al. 1994 consensus conference on acute GVHD grading. Bone Marrow Transplant. 1995;15:825-828.)
Time Frame: Within 100 Days Post-SCT (Stem Cell Transplant)
Measure: Count of Participants; unit: Participants
Groups:
- Cohort B- Related Donor- Dose Level 1: Dose Level 2 of Clofarabine will be administered 52 mg/m2/dose Day -6 through -2. Cohort B will include patients who have matched related donors.
- Cohort C- Unrelated Donor- Dose Level 2: Dose Level 1 is the starting dose level of Clofarabine will be 40 mg/m2/dose given day -6 through -2. A modified 3+3 patient cohort dose escalation and de-escalation design. Cohort C will include patients who have unrelated donors.
Arm/Group | Cohort A- Related Donor- Dose Level 1 | Cohort B- Related Donor- Dose Level 1 | Cohort C- Unrelated Donor- Dose Level 2 | Cohort D- Unrelated Donor- Dose Level 2
Number analyzed (Participants) | 3 | 6 | 3 | 6
Participants | 1 | 3 | 1 | 3

6. Post Hoc Outcome: CD3 Donor Chimerism at Day 30 (Full Donor)
Description: Donor engraftment was assessed by testing of chimerism in the T cell (CD3) subpopulation at day +30 done by local institution using PCR-based analyses of polymorphic microsatellite regions.
Time Frame: Day 30
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A- Related Donor- Dose Level 1 | Cohort B- Related Donor- Dose Level 2 | Cohort C- Unrelated Donor- Dose Level 1 | Cohort D- Unrelated Donor- Dose Level 2
Number analyzed (Participants) | 3 | 5 | 3 | 6
Participants | 2 | 4 | 3 | 6

7. Post Hoc Outcome: CD3 Donor Chimerism at Day 30 (Mixed Chimerism)
Description: as for outcome 6
Time Frame: Day 30
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A- Related Donor- Dose Level 1 | Cohort B- Related Donor- Dose Level 2 | Cohort C- Unrelated Donor- Dose Level 1 | Cohort D- Unrelated Donor- Dose Level 2
Number analyzed (Participants) | 3 | 5 | 3 | 6
Participants | 1 | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: 3 years, 1 month
Description: The definitions of AE and SAE do not differ from the clinicaltrials.gov definitions
Groups:
- 40 mg/m2 Dose: Patients who received the starting dose level of 40 mg/m2
- 52 mg/m2 Dose: Patients who received the increased dose level of 52 mg/m2
Arm/Group | 40 mg/m2 Dose | 52 mg/m2 Dose
All-Cause Mortality (participants affected / at risk) | 1/6 | 5/12
Serious Adverse Events (participants affected / at risk) | 1/6 | 0/12
Other Adverse Events (participants affected / at risk) | 6/6 | 10/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 40 mg/m2 Dose (N=6) | 52 mg/m2 Dose (N=12)
Fever (General disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 40 mg/m2 Dose (N=6) | 52 mg/m2 Dose (N=12)
Abdominal pain NOS (Gastrointestinal disorders) | 0 | 1
Adrenal insufficiency NOS (Endocrine disorders) | 0 | 1
Alanine aminotransferase increased (Investigations) | 6 | 4
Anorexia (Metabolism and nutrition disorders) | 2 | 5
Aspartate aminotransferase increased (Investigations) | 5 | 3
Dehydration (Gastrointestinal disorders) | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 1 | 0
Dermatitis exfoliative NOS (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatology-Other (Skin and subcutaneous tissue disorders) | 1 | 1
Diarrhea NOS (Gastrointestinal disorders) | 0 | 1
Hemoglobin (Blood and lymphatic system disorders) | 1 | 3
Hemoglobinuria (Blood and lymphatic system disorders) | 1 | 0
Hyperglycemia NOS (Metabolism and nutrition disorders) | 0 | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycemia NOS (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 2
Hypotension NOS (Vascular disorders) | 0 | 1
Infection w/ Gr 3/4 ANC, Blood (Infections and infestations) | 1 | 0
Infection w/ norm ANC, Catheter (Infections and infestations) | 0 | 1
Infection w/ norm ANC, Colon (Infections and infestations) | 0 | 1
Infection-Other (Infections and infestations) | 0 | 1
Leukopenia NOS (Blood and lymphatic system disorders) | 3 | 5
Lymphopenia (Blood and lymphatic system disorders) | 2 | 5
Metabolic/Lab-Other (Metabolism and nutrition disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 2
Neutrophil count (Blood and lymphatic system disorders) | 3 | 5
Pain - Other (General disorders) | 0 | 1
Platelet count decreased (Blood and lymphatic system disorders) | 2 | 7
Syncope (Nervous system disorders) | 0 | 2
Vision blurred (Eye disorders) | 0 | 1
Vomiting NOS (Gastrointestinal disorders) | 0 | 1
Weight increased (Metabolism and nutrition disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days